CLINICAL TRIAL: NCT01206634
Title: Effect of Regenerative Injection Therapy on Function and Pain in Patients With Knee Osteoarthritis
Brief Title: Regenerative Injection Therapy and Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Responsible Party: Dr Richard Dumais, anastesiologist, Réseau de Santé Vitalité Health Network
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HC-9427-B2716-21C
Record Dates: First submitted 2010-09-17; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Knee Arthrosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regenerative injection therapy (Experimental)
  Interventions: Procedure: Regenerative injection therapy
- Exercise (Active Comparator)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Procedure: Regenerative injection therapy — Injections of 1cc of a 15% dextrose and 0.6% lidocaine solution free of adrenaline in each of eight administration sites in the collateral ligaments and a 5 cc injection of a 20% dextrose and 0.5% lidocaine without adrenaline solution inside the knee joint.
  Arms: Regenerative injection therapy
Behavioral: Exercise — the exercise program consists of 4 strengthening exercises for which participants are asked to perform 3 sets of 10 repetitions daily
  Arms: Exercise

SUMMARY:
The objective is to assess the effectiveness of regenerative injection therapy (RIT) to relieve pain and restore function in patients with knee osteoarthritis.

The study design is a randomized controlled trial with cross-over. 40 patients with chronic knee osteoarthritis will be randomly assigned to receive exercise therapy for 32 weeks in combination with RIT on weeks 0, 4, 8, and 12 or exercise therapy for 32 weeks combined to RIT on weeks 20, 24, 28 and 32. The primary outcome is the WOMAC score.

DETAILED DESCRIPTION:
The administration of treatment as used in this study was approved by Health Canada and the study received ethical approbation by the regional health authority Institutional Review Board. Health Canada number: 9427-B2716-21C.

Participants meeting will be randomized into one of two study groups using opaque sealed envelopes in blocks of 6. Each envelope contains a description of the intervention of assignment. For group A, the intervention consists of a conventional physiotherapist supervised exercise program for 32 weeks in combination with RIT on weeks 0, 4, 8, and 12. Intervention for group B includes the supervised exercise program for 32 weeks in combination with RIT on weeks 20, 24, 28 and 32 of follow-up. For all study participants, the exercise program consists of 4 strengthening exercises for which participants will be asked to perform 3 sets of 10 repetitions daily.

RIT injections: The osteo-tendinous junction of both insertion sites of the collateral ligaments will be identified. Patients will then receive injections of 1cc of a 15% dextrose and 0.6% lidocaine solution free of adrenaline in each of eight administration sites in the collateral ligaments. A 5 cc injection of a 20% dextrose and 0.5% lidocaine without adrenaline solution will also be administered inside the knee joint. The intra-articular injection will be performed using the anterior approach. Solutions are prepared by a hospital pharmacist the morning of the injections. Each infiltration will be preceded by a local sterilization consisting of three disinfections with a 2% chlorexidine and 4% idopropyl alcohol solution.

Study variables Several measures of functional capacity and pain are used. The primary outcome is the Western Ontario and McMaster Universities Osteoarthritis Index of severity of osteoarthrosis symptoms (WOMAC version 3.1). This self-administered questionnaire assesses pain, disability and joint stiffness using 24 items with 5-point Likert scales. Other outcomes included the Brief Pain Inventory (short form), which is administered to assess pain intensity and pain-related functional impairment (physical and emotional). More specifically, four items assess the intensity of current pain and pain at its least, worst, and average during the past day on scales from 0 ("no pain") to 10 ("pain as bad as you can imagine"). Seven more items measure pain-related functional interference in different domains (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life) rated from 0 ("does not interfere") to 10 ("interferes completely"). Participants will also rate their pain with the Wong-Baker Faces Pain Rating Scale, a series of 6 faces anchored at 0 for "no hurt" and 5 for "hurts worst". After being instructed that each face is for a person who feels happy because he has no pain or sad because he has some or a lot of pain, participants chose the face that best describes how they feel. Participants also rate their pain with a simple descriptive intensity scale with 7 adjectives (no pain, mild pain, moderate pain, severe pain, very severe pain, and worst pain possible), a numeric distress scale with anchors 0 for "no pain" and 10 for "unbearable pain", and a visual analogue scale with the words "no pain" and "pain as bad as could possibly be" at the left and right ends of the line, respectively. The Timed Up-and-Go Test will be used to evaluate functional capacity. Participants start in a sitting position (with hands resting on the arms of an armchair of standard height), stand up, walke 3 meters, turn around, and walk back to sit down on the chair again. The timing starts when the participant's back comes off the chair, and stops when their buttocks touch the seat of the chair.

Patients' severity of knee osteoarthritis will be assessed by a radiologist using the Kellgren-Lawrence grading scale. Anteroposterior radiographs of the knee are to be taken prior to enrollment in the study.

Follow up Participants will meet with research assistants (research nurses and family medicine residents) at the onset of the study, every four weeks of the subsequent 32 weeks of intervention, and four weeks after the intervention. At each of those visits, participants will be asked to fill in measurement questionnaires. Research assistants will also investigate the presence of side effects or complications and remind participants that the research protocol restricts them from taking any anti-inflammatory medication throughout the 32 weeks of intervention. Participants will also meet the physiotherapist every four weeks to review exercises. At the onset of the study, participants will receive a study calendar detailing each of their appointments. In addition, patients will receive an appointment card at the end of each visit. This card provides the time of the next visit, contact information, as well as a list of conditions for which participants should contact the study center. If a participant presents a sustained deterioration of symptoms or function, or experiences undesirable side effects, the presumed contributing part of the treatment will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* have had a diagnosis of knee arthrosis,
* experience pain in the knee for a minimum of six months,
* be capable to understand and execute physiotherapy exercises,
* be 18 years or older.

Exclusion Criteria:

* previous operation of the referring knee,
* infection of the skin surrounding the knee or of the articulation,
* abnormal coagulation,
* allergy to lidocaine,
* pregnancy,
* breast feeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index of severity of osteoarthrosis symptoms (WOMAC version 3.1) | Every 4 weeks from week 0 to 36
  This self-administered questionnaire assesses pain, disability and joint stiffness using 24 items with 5-point Likert scales.

SECONDARY OUTCOMES:
Brief Pain Inventory (short form) | Every 4 weeks from week 0 to 36.
Wong-Baker Faces Pain Rating Scale | Every 4 weeks from week 0 to 36.
Timed Up-and-Go Test | Every 4 weeks from week 0 to 36.
  Measure of patients mobility. Patients start sitting on a chair, they then stand, walk a short distance, turn around, and come back to sit on the chair again. Score = Time to complete the task.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dumais, MD, Principal Investigator — Dr. Georges-L.-Dumont Regional Hospital, Vitalité Health Network